CLINICAL TRIAL: NCT04841447
Title: Tumor Cell and DNA Detection in the Peripheral Blood of Patients With Hematological Malignancy
Brief Title: Membrane Target Detection for Leukemia Treatment
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Xunlei Kang, Associate Professor, University of Missouri-Columbia
Other Study IDs: 2018932
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Study sample collection — Peripheral blood draws and bone marrow aspiration will be done during clinic visit and hospital stay.

SUMMARY:
Acute myeloid leukemia (AML) accounts for more than 40% of leukemia mortality in the United States. Each year around ten thousand people die from the disease, most within a few years of diagnosis. Despite advances in our understanding of the disease, few improvements in the therapy of AML have been made. Collecting specimens from the blood and bone marrow will increase understanding of the effect of Dipeptidyl Peptidase-4 (DPP-4) Inhibitors on human AML-SCP to develop individualized therapies. We also found DPP4 is highly expressed in other hematological malignancies in our mouse model, thus we would like to use human samples to investigate the role of DPP4 in hematological malignancy development and the mechanism underlying, especially to deeply understand the role of DDP4 in leukemia.

DETAILED DESCRIPTION:
Specific targets and novel strategies to eliminate AML stem cells are required for AML treatment. Collecting specimens from the blood and bone marrow will increase understanding of the effect of DPP4 inhibitors on human AML-SCP to develop individualized therapies. We will test the effect of DPP4 inhibitors on human AML-SCP in vitro and in vivo and whether the addition of DPP4 inhibitors can prevent AML relapse once the disease is in the remission stage.

Chronic myeloid leukemia (CML) is a stem cell (SC) neoplasm characterized by the BCR/ABL1 oncogene. CML is a steadily developing blood and bone marrow disease that has three stages: chronic, accelerated, and blastic. If it reaches the blastic process, it is known as acute leukemia, which is the same as AML. While the mechanisms of BCR/ABL1-induced transformation are well understood, little is known about the effector molecules that contribute to leukemic SC (LSC) malignant expansion and extramedullary spread in CML. Furthermore, DPP4 is not only highly expressed in leukemia samples, but also specifically expressed in some of the other hematological malignancies, such as AML, CML, ALL, CLL, Lymphomas, or Myelomas, and may work as a stem cell marker as well. At this point, we would like to use human blood samples to investigate the role of DPP4 in hematological malignancy to deeply understand the role of DPP4 in leukemia.

ELIGIBILITY:
Inclusion Criteria:

* All hematological malignancy patients.
* Must be 18 years old.

Exclusion Criteria:

* Participants with impaired decision-making capacities;
* Pregnant women or fetuses;
* Children (under 18 in Missouri, also dependent on State law);
* Non-viable neonates or neonates of uncertain viability (neonates=newborns);
* Non-English-speaking subjects;
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hematological malignancy patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
DPP4 inhibitors measured in blood samples will be correlated with patient survival data. | 5 years
  DPP4 inhibitors measured in blood samples will be used in vitro and in vivo a pre-clinical model.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No